CLINICAL TRIAL: NCT06385288
Title: Blood and Tissue Extraction for Immunological Examinations During Neoadjuvant Therapy of Soft Tissue Sarcomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 268/2021BO2
Record Dates: First submitted 2023-11-23; First posted 2024-04-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Soft Tissue Sarcoma Adult
Keywords: Soft tissue sarcomas; immunological examinations; neoadjuvant therapy; radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Blood Specimen Collection; Tissue Banks; Neoadjuvant Therapy

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm trial (Other): Blood and tissue collection for immunological studies under neoadjuvant Therapy of soft tissue sarcomas. Prospective data collection and translational accompanying research on standard therapy. Use of tissue, blood samples and advanced imaging.
  Interventions: Other: Blood and tissue collection for immunological studies, advanced imaging.; Other: neoadjuvant Therapy

INTERVENTIONS:
Other: Blood and tissue collection for immunological studies, advanced imaging. — Blood and tissue collection for immunological studies under neoadjuvant Therapy of soft tissue sarcomas. Prospective data collection and translational accompanying research on standard therapy. Use of tissue, blood samples and advanced imaging.
Other: neoadjuvant Therapy — neoadjuvant Therapy

SUMMARY:
"Blood and Tissue Extraction for Immunological Examinations During Neoadjuvant Therapy of Soft Tissue Sarcoma" is a prospective study with additional translational research using preoperative and postoperative tissue, blood sampling and advanced imaging.

DETAILED DESCRIPTION:
All patients (> 18 Years) with histologically confirmed high-risk soft tissue sarcoma eligible for neoadjuvant multimodal therapy (including radiotherapy +/- concomitant and sequential chemotherapy +/- hyperthermia as well as surgery) are screened for the study. Neoadjuvant therapy consists of 50-50.4 Gy in 25-28 fractions. Additional concomitant or sequential chemotherapy may be applied in selected cases (young patients, high-grade tumors). Additional hyperthermia concomitant to neoadjuvant radiotherapy is applied in selected cases if not contraindicated.

Preoperative tissue sampling to generate primary tumor cell lines in additional translational research is performed in each patient with a lesion suspect for soft tissue sarcoma and eligible for multimodal therapy. Primary cell lines are analyzed biologically (growth pattern, radioresistance, migration, molecular markers RT-PCR, immunological properties such as immunogenic cell death, lysis by cellular immunotherapies such as CAR-NK cells. Postoperative tumor tissues are additionally analyzed for immune cell mapping using complex immunohistochemistry. Biopsy and resection should include proteome analysis and DNA sequencing (only of the tumor tissue, not normal tissue).

Additional immunological monitoring (including cellular immune status, serum marker e.g. cell free DNA, HMGB1) is performed using blood sampling with in total 4 blood controls (25 ml each, before neoadjuvant radiotherapy, during the second and last week of radiotherapy as well as before surgery). In patients treated with concomitant MR-guided hyperthermia, weekly MR-imagine is performed.

Follow-up is carried out as part of the oncological controls over 5 years. The overall study is planned over a period of 5 years (interventional part), additional 5 years follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Planned histological confirmation for especially high-risk soft tissue sarcoma via open Sampling
* Indication for neoadjuvant multimodal therapy (radiation and locoregional Hyperthermia, optionally with simultaneous chemotherapy)
* Planned resection of a department of the CWS
* Age > 18 years
* Ability to consent
* Additionally for imaging study: Treatment on the combined MR hyperthermia device

Exclusion Criteria:

* Age < 18 years
* Poor understanding (language etc.)
* Lack of reconnaissance ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2031-07-21 (Estimated)

PRIMARY OUTCOMES:
Description of the cellular immune status via flow-cytometrie from collected blood samples | 5 years of recruitment, 5 years follow-up
  Blood samples are taken on the days of simulation-CT, first and third week of the radiation therapy, as well as before surgery.
Description of the cellular immune status on tissue samples ussing komplex immunohistochemie | 5 years of recruitment, 5 years follow-up
  Tissue samples are taken as incisional biopsie as well as in the tumor tissue after the surgery
Measurement of the cellular free DNA from collected blood samples | 5 years of recruitment, 5 years follow-up
  Blood samples are taken on the days of simulation-CT, first and third week of the radiation therapy, as well as before surgery.
Measurement of HMGB1 from collected blood samples | 5 years of recruitment, 5 years follow-up
  Blood samples are taken on the days of simulation-CT, first and third week of the radiation therapy, as well as before surgery.
Evaluation of morphological tumor characteristics (size, diffusion) with weekly MRIs | 5 years of recruitment, 5 years follow-up
  Weekly MRIs during neoadjuvant radiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No